CLINICAL TRIAL: NCT05010577
Title: A Phase 1b/2a, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Nebulized Bacteriophage Treatment in Outpatient Adult Cystic Fibrosis (CF) Subjects With Chronic Pseudomonas Aeruginosa (PsA) Pulmonary Infection
Brief Title: Nebulized Bacteriophage Therapy in Cystic Fibrosis Patients With Chronic Pseudomonas Aeruginosa Pulmonary Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BiomX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMX-04-001
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pseudomonas Aeruginosa Infection; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BX004-A (Experimental): Participants will be randomized to receive standard dose of nebulized bacteriophage
  Interventions: Drug: BX004-A
- Placebo (Placebo Comparator): Participants will be randomized to receive nebulized placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BX004-A — Combination of nebulized bacteriophages targeting Pseudomonas aeruginosa
  Other Names: Bacteriophage
  Arms: BX004-A
Drug: Placebo — Nebulized placebo
  Other Names: Vehicle buffer
  Arms: Placebo

SUMMARY:
This is a Phase 1b/2a study with the primary objective to determine if BX004-A is safe and tolerable. Exploratory objectives include whether BX004-A reduces sputum Pseudomonas aeruginosa (PsA) bacterial load in CF subjects with chronic PsA pulmonary infection.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter study to evaluate the safety and tolerability of BX004-A in CF subjects with chronic PsA pulmonary infection. The study is divided into two parts, a single-ascending and multiple-dose phase (Part 1) and a multiple dose phase (Part 2). Subjects in both parts will be included in a 6-month safety follow-up. A Data Safety Monitoring Board will monitor safety in both parts. The purpose of the study is to evaluate safety and tolerability of BX004-A, and whether BX004-A reduces the PsA burden in the sputum of CF subjects with chronic PsA pulmonary infection. Clinically stable CF subjects with a confirmed diagnosis of CF and chronic PsA pulmonary infection will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Cystic fibrosis patients with chronic Pseudomonas aeruginosa pulmonary infection receiving standard of care CF medications
* Age ≥ 18 years
* FEV1 ≥ 40% predicted
* Clinically stable lung disease
* Willing and able to provide adequate sputum samples, using any method (spontaneously expectorated, induced, from home or clinic) at designated study visits.

Key Exclusion Criteria:

* Known hypersensitivity to bacteriophages or excipients in the formulation.
* Receipt of prior bacteriophage therapy within the 6 months prior to Screening
* Recovery of Burkholderia species from respiratory tract within 1 year prior to screening
* Currently receiving treatment for allergic bronchopulmonary aspergillosis
* Currently receiving treatment for active infection with non-tuberculous mycobacteria
* History of severe neutropenia
* History of lung transplant
* History of solid organ transplant
* Acquired or primary immunodeficiency syndrome
* Initiation or change in CF modulator therapy less than 3 months prior to screening
* Pregnant or breastfeeding female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months
  Incidence of treatment emergent adverse events following single and multiple doses of BX004-A administered by inhalation

OTHER OUTCOMES:
PsA burden in sputum at various timepoints | 1 month
  Change in PsA colony-forming units (CFU) per gram of sputum

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — BiomX, Inc.
Locations (28):
- United States (18):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - New York Medical College, Valhalla, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University Hospitals Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Texas Children Clinic, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- University Hospital in Motol, Prague, Czechia
- Israel (5):
  - Rambam Health Care Campus (RHCC) - Ruth Rappaport Children's Hospital, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah University Medical Center, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tikvah
  - The Chaim Sheba Medical Center, Ramat Gan
- Netherlands (2):
  - Amsterdam Medical Center, Amsterdam
  - University Medical Center Utrecht, Utrecht
- Spain (2):
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Vall d'Hebron Barcelona Hospital Campus, Barcelona

IPD SHARING:
Plan to Share IPD: No